CLINICAL TRIAL: NCT03133598
Title: Prospective Cohort Study of Interventional Therapy and Craniotomy for Unruptured Aneurysms
Brief Title: Treatment of Unruptured Intracranial Aneurysms in China
Status: Completed | Type: Observational
Sponsor: Zhujiang Hospital (Other)
Collaborators: Xuanwu Hospital, Beijing (Other); Beijing Tiantan Hospital (Other); Guangdong Provincial People's Hospital (Other); First Affiliated Hospital of Chongqing Medical University (Other); The Affiliated Hospital Of Southwest Medical University (Other); West China Hospital (Other); Shenzhen Second People's Hospital (Other); Guangdong 999 Brain Hospital (Other); Shantou Central Hospital (Other); ZhuHai Hospital (Other); Zhongshan Hospital Of Traditional Chinese Medicine (Other); Third Affiliated Hospital, Sun Yat-Sen University (Other); Eighth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Duan Chuanzhi, Deputy director, department of neurosurgery, southern medical university, Guangzhou, Zhujiang Hospital
Other Study IDs: 2016YFC1300804
Record Dates: First submitted 2017-04-07; First posted 2017-04-28 (Actual); Last update posted 2024-09-23 (Actual); Status verified 2024-09

CONDITIONS: Intracranial Aneurysm; Stent Embolisation; Craniotomy; Coil-assissted Embolisation; Covered Stent; Woven EndoBridge
Keywords: Un-ruptured intracranial aneurysm; Interventional therapy and craniotomy; Prospective cohort study; China
MeSH Terms: conditions — Intracranial Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- 1: patients with intracranial aneurysms who underwent endovascular or miro-neurosurgical treatment

SUMMARY:
Un-ruptured intracranial aneurysm is a complex disease that seriously affects human life and health. At present, the treatment of intracranial aneurysm is divided into interventional treatment and craniotomy clipping, the two treatment methods are different in the intervention effect of aneurysm, for example, the complications of interventional therapy are lower than craniotomy clipping, but the long-term patency rate is lower than craniotomy clipping, and there is no standard of treatment in different parts of aneurysm in our country, the choice of intervention measures of un-ruptured aneurysm is different in different clinical centers; on the other hand, there are serious problems in the treatment of aneurysms, because without the relevant guidelines of diagnosis and treatment of intracranial aneurysms, different clinical centers will cause excessive treatment of un-ruptured aneurysms, not only bring unreasonable utilization of medical resources, but also cause the subject's life and property to be threatened.

The patients with un-ruptured intracranial aneurysm(estimated sample number over 1500) were included in prospective cohort study, after clipping and intervention operation, setting fixed time for postoperative follow-up, the clinical data and image data were recorded, the safety, efficacy and economic benefits of interventional treatment and craniotomy clipping were compared, providing strategies for the standardized treatment of un-ruptured intracranial aneurysms.

DETAILED DESCRIPTION:
For this study,investigators consulted and hired professionals and experts about data collection, data and methodology,including Data Monitoring Committee, Data Management Committee, Progect Academic Committee, Executive Group, Project Manager, Project Statistician,Technical Support Center. investigators have a scientific regulations for this project. Project Manager and Executive Group: To ensure the successfully implementation of this project, including charging the daily operations of the study in 20 different research hospitals, organizing the monthly meeting to consider issures raised during the monthly progress of the study, liaising with the steering committee,the data management centre and statistical centre. Data management Committee: To be responsible for setting up and maintain the Electronic Data Capture (EDC) System according to the papera Case Report Form(pCRF) designed by principal investigators. To collect and save the pCRF coming from sub-centers. To entry the data into EDC system and keep the same with CRF. To organize training for the investigators about the rules in filling the EDC and pCRF.To determine the frequency of the Data Management Report and to fed it back to the steering committee every three months. Data Mornitoring Committee: To determine the frequency of the data mornitoring including the source data(Medical records) accuracy, completeness and representativeness comparing the external data(EDC, pCRF) in participanted centers.

To report the results after the mornitoring back to the steering committee about the missing data, non-reported and other problems about the study. To make a Standard Operation Procedure(SOP) from getting data to using data. Academic Committee: To supervise the academic issues including patient recruitment, protocol deviation, adverse events evalutating. To settle down the question and problem in the process of the study. Project Statistician: We cooperate with the statisticians of Medical Research & Biometrics Center National Center for Cardiovascular Diseases, China to get the perfessional statistical report. Technical Support Center:To provide technical support during the process of the study.

ELIGIBILITY:
Inclusion Criteria:

1. At least one imaging methods( CTA / MRA / DSA ) confirmed un-ruptured intracranial aneurysms, whether have clinical symptoms or not;
2. For multiple aneurysms, regardless of previous treatment, the requirement for treatment interval should > 6 months.
3. The patient has the autonomous life ability, the scores of MRS≤ 3 points;
4. The subjects age > 14 years
5. subjects or family members agree to sign informed consent.

Exclusion Criteria:

1. Intracranial aneurysms and with 30 days of unexplained subarachnoid hemorrhage;
2. Subjects with other intracranial vascular malformations, such as AVM, AVF, etc.;
3. Subjects with malignant tumors in the intracranial or other parts of the body;
4. Fusiform, traumatic, bacterial or dissecting aneurysm;
5. Subjects with severe mental illness unable to communicate when diagnosing disease;
6. The body condition is poor, the survival time is less than 1 year or poor physical condition, can not tolerate the general anesthesia or aneurysm surgery;
7. Subjects involved in other intracranial aneurysms related clinical research;
8. A patient who received surgical clipping or endovascular treatment at once;
9. Subjects who were not followed up.
10. < 3 mm intracranial aneurysm。

Ages: 14 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with un-ruptured intracranial aneurysms.
Sampling Method: Non-Probability Sample
Enrollment: 5126 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2022-12-30 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The safety evaluation of interventional therapy and craniotomy clipping. | 6 months later after operation.
  The safety evaluation including the mortality（mRS=6） rate and disability（2<mRS<6） rate of subjects.
The effectiveness evaluation of interventional treatment . | 6 months later after operation.
  The effectiveness evaluation including the complete occlusion（Raymond classification=1） rate of aneurysms.
Clinical function prognosis | 1 year
  0 completely silent
  1. despite symptoms, but not visibly disabled, can complete all regular duties and activities
  2. mild disabilities, not all activities previously possible, but can deal with personal affairs without need of assistance
  3. moderate disability requires some help, but walking does not need assistance
  4. severe disabilities, unable to walk independently, no others can not meet their needs
  5. severely disabled, bedridden, Urine, requiring continuous care and care
  6. mortality
Raymond classification | 1 year
  1. Complete occlusion
  2. Partial occlusion
  3. Recurrence
The effectiveness evaluation of craniotomy clipping. | 6 months later after operation.
  The effectiveness evaluation including the recurrence（Raymond classification=3） rate of aneurysms.

SECONDARY OUTCOMES:
The safety evaluation of interventional therapy or craniotomy clipping. | up to 24 months
  The safety evaluation including the mortality（mRS=6） rate and disability（2<mRS<6） rate of subjects.
The effectiveness evaluation of interventional treatment or craniotomy clipping. | up to 24 months
  The effectiveness evaluation including the complete occlusion（Raymond classification=1） rate of aneurysms.
The success rate of treatment or craniotomy clipping. | up to 24 months
  angiography revealed total or near total occlusion of aneurysm in 6 months after operation, no recurrence of aneurysm was found, the treatment was considered successful.
The incidence of major adverse events during follow-up. | up to 24 months
  cerebrovascular complications including any intracranial hemorrhage, ischemia, or death
The cost of interventional therapy or craniotomy clipping. | up to 24 months
  All costs associated with treatment

CONTACTS AND LOCATIONS:
Overall Officials: Chuanzhi Duan, Ph.D., Principal Investigator — Department of Neurosurgery, Southern Medical University, Zhujiang Hospital
Locations (1):
- Southern Medical University, Zhujiang Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
Data are available upon reasonable request. The data supporting this study's findings are available from the Principal Investigator （Chuanzhi Duan） upon reasonable request.

REFERENCES:
- [Derived] Chen Y, Fan H, He X, Guo S, Li X, He M, Qu Y, Yang X, Zhang H, Sun X, Wang L, Wang Z, Tong X, Zhong M, Maimaitili A, Tong Z, Duan C. China Intracranial Aneurysm Project (CIAP): protocol for a prospective cohort study of interventional treatment and craniotomy for unruptured aneurysms. BMJ Open. 2018 May 24;8(5):e019333. doi: 10.1136/bmjopen-2017-019333. PMID 29794089